CLINICAL TRIAL: NCT03572335
Title: Systems Biology of Diffusion Impairment in HIV--BoDI
Brief Title: Systems Biology of Diffusion Impairment in Human Immunodeficiency Virus (HIV)
Acronym: BoDI
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Alison Morris, Professor of Medicine, University of Pittsburgh
Other Study IDs: STUDY19050326
Record Dates: First submitted 2018-06-13; First posted 2018-06-28 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-08

CONDITIONS: HIV Infections; Pulmonary Disease
Keywords: HIV; emphysema; diffusing capacity; chronic obstructive pulmonary disease(COPD)
MeSH Terms: conditions — HIV Infections; Lung Diseases; Emphysema; Pulmonary Disease, Chronic Obstructive | interventions — Respiratory Function Tests; Walk Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, saliva, oral wash, stool
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- HIV positive with normal PFT's: HIV positive with normal baseline DLco. Subjects with DLco>80% predicted after adjustments for Hgb and Co
  Interventions: Diagnostic Test: PFT's (pulmonary function testing)
- HIV positive with mild DLco impairment: HIV positive with mild DLco impairment DLco <80% predicted after adjustments for Hgb and Co.
  Interventions: Diagnostic Test: PFT's (pulmonary function testing)

INTERVENTIONS:
Diagnostic Test: PFT's (pulmonary function testing) — The routine lung function endpoints of FVC(forced vital capacity), FEV1, FEV1/FVC, and FEF25-75% will be measured with the flow-volume loop recorder before and after bronchodilator administration. The system is calibrated for body temperature and pressure of saturated gas and volumes, per American Thoracic Society (ATS) standards . DLco will be measured using the automated single-breath procedure of the integrated testing system, which conforms with ATS standards.
  Other Names: 6MWT (6 minute walk test)

SUMMARY:
Diffusing capacity for carbon monoxide (DLco) abnormalities are common in HIV+ individuals and associated with significant morbidity and mortality. The complexity and the individualized differences in causes of these abnormalities have been challenging to unravel using traditional approaches. In this proposal, the investigators construct a systems' modeling approach to identify novel molecular and clinical pathways contributing to DLco impairment in HIV+ individuals and to determine predictive signatures of DLco decline in order to develop strategies to treat and prevent abnormal lung function in this susceptible population.

DETAILED DESCRIPTION:
Mechanisms of impairment of diffusing capacity for carbon monoxide (DLco), which affects over 50 percent of HIV+ individuals, are poorly understood. No therapies exist despite significant impact on quality of life and mortality. Identifying molecular pathways of DLco impairment in HIV+ individuals and developing ability to predict HIV+ individuals at risk of DLco impairment is thus of utmost importance for improving care. In this proposal, the investigators construct a systems' modeling approach to identify molecular and clinical pathways contributing to DLco impairment in HIV+ individuals. The investigators collect multiple parallel molecular datasets integrated with detailed pulmonary function, radiographic, and echocardiographic measurements to build a comprehensive, systems level model of DLco abnormalities in HIV and to develop predictive models of susceptibility to DLco worsening. As our preliminary data suggest that certain micro ribonucleic acid (miRNAs), such as the hypoxia-induced and metabolically active gene (miR-210), may play an important role in DLco abnormalities in HIV, the investigators then perform hypothesis-testing experiments to determine the impact of miRNAs on lung epithelial and endothelial cells. The investigators will utilize a well phenotyped cohort of over 500 HIV+ individuals with associated biospecimens to execute the aims.

Participants identified to already have specimens available will be scheduled to have PFT testing, bronchoscopy including bronchial wash with brushes and blood collection.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age 18 to 80
2. HIV positive and participated in previous HLRC(HIV Lung Research Center) study (PRO10060177, PRO09050521, PRO14070355, PRO08030011, PRO00606151, PRO13050229, PRO17060077).
3. Negative pregnancy test (for women of child barring capabilities).
4. Have undergone bronchoscopy with BAL(bronchial lavage) and/or brushing for AECs in storage.
5. Receiving ART (Anti-Retroviral Therapy)and virally-suppressed for at least 6 months.

Exclusion Criteria:

1. Pregnancy or breast-feeding. (urine pregnancy done on all females of child bearing potential-males and females who are at least 1 year post menopausal or surgically sterile will not be tested)
2. Contraindication to pulmonary function testing (i.e. abdominal or cataract surgery within 3 months, recent myocardial infarction, etc.).
3. Increasing respiratory symptoms or febrile (temperature >100.40F [380C]) within 4 weeks of study entry.
4. Acute cardiopulmonary issue in the past 4 months.
5. Uncontrolled hypertension at screening visit (systolic > 180 mm Hg or diastolic > 100 mm Hg) from an average of two or more readings. Subject may return for screening after blood pressure is controlled.
6. Active cancer requiring systemic chemotherapy or radiation.
7. Active infection of lungs, brain, or abdomen.
8. Intravenous drug use or alcohol use that will impair ability to complete study investigations in the opinion of the investigator.
9. subjects with an upper or lower respiratory tract infection
10. individuals receiving chronic or acute antibiotics in the prior 4 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18-80 year old men and women who are HIV positive. All will be pulled from previous HIV/Lung studies done by the same PI
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Identify key causal molecular pathways of DLco impairment. | 3 years
  elucidating complex associations and causal relationships between clinical characteristics, the host inflammatory response, cellular metabolism, the microbiome, and miRNAs.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Morris, MD, MS, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh department of medicine division of Pulmonary, Allergy and Critical Care medicine, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No